CLINICAL TRIAL: NCT05300646
Title: The Effect of an Adapted Mindfulness-Based Stress Reduction Program on Mental Health, Maternal Bonding and Birth Outcomes in Psycho-socially Vulnerable Pregnant Women: a Randomized Controlled Trial.
Brief Title: Mindfulness-Based Stress Reduction for Psycho-socially Vulnerable Pregnant Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2554
Record Dates: First submitted 2022-03-10; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Perinatal Mental Health; Pregnancy Related
Keywords: Mindfulness; Mindfulness-based stress reduktion; MBSR; Perinatal mental health; Self-compassion

STUDY DESIGN:
Intervention Model Description: A single-center, parallel group, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Group affiliation will be concealed for the researcher performing the statistical analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The prenatal MBSR program is an adaptation of MBSR. Details on the adaptation process is described in Skovbjerg S et al. Pilot and feasibility studies, 2021 Jun 3; 7 (1):118. Prenatal MBSR include nine weekly two-hour classes and is delivered in a combination between physical attendance and live-online teaching. The recommended time for daily mindfulness training between sessions is 15 minutes a day with options for longer practice. Audio recordings with guided meditations and a video with yoga programs for pregnancy is provided for home practice.
  Interventions: Behavioral: Prenatal mindfulness-based stress reduction
- Treatment as usual (No Intervention): Standard clinical practice, usual care (TAU), consists of an average of six routine pregnancy visits to the outpatient antenatal clinic at Copenhagen University Hospital, Hvidovre and to a General Practitioner. Routine pregnancy visits involves primarily preventive counselling by midwifes, and in some cases consultations with a physician or social worker throughout pregnancy and the early post-partum period. In some cases, usual care may include consultations with a psychologist, although usually limited to a few sessions, and in more severe cases referral to psychiatric treatment.

INTERVENTIONS:
Behavioral: Prenatal mindfulness-based stress reduction — An adapted mindfulness-based stress reduction (MBSR) program with a particular focus on pregnancy and early motherhood.
  Arms: Intervention

SUMMARY:
The aim of the study is to address the need for a wider array of evidence-based and non-pharmacological options to improve mental health in a psycho-socially highly vulnerable group of pregnant women. In more detail, the primary outcome is to estimate the effect of prenatal Mindfulness-Based Stress Reduction (MBSR) as an add-on to usual care on mental well-being when compared to usual care alone. Second, to estimate the effect of prenatal MBSR on perceived stress and symptoms of depression and anxiety, and third to explore the effect on maternal bonding and childbirth, e.g. gestational age and experience of childbirth. Finally, to examine the mediating effect of mindfulness and self-compassion on the primary outcome.

DETAILED DESCRIPTION:
Background A history of psychopathology or psychosocial adversities are risk factors for mental disorders in the perinatal period. Mental disorders in pregnancy can adversely affect the developing fetus, which call for early prevention. Mindfulness-Based-Stress-Reduction (MBSR) is an acceptable intervention for pregnant women and has a growing evidence-base with meta-analyses consistently pointing to reductions in symptoms of stress, anxiety and depression. The aim of this study is to address the need for a wider array of evidence-based and non-pharmacological options to improve mental health in a psychosocially highly vulnerable group of pregnant women.

Methods/design Pregnant women (n = 238) referred to an outpatient clinic at Copenhagen University Hospital, Amager and Hvidovre, Denmark will be recruited for the study. The design is a single-center, parallel group, randomized controlled trial, with an adapted MBSR program as add on to usual care. The primary outcome is mental wellbeing. Secondary and exploratory outcomes include stress, anxiety, depression, mindfulness, compassion, antenatal attachment and childbirth experience. Participants will be randomized in a 1:1 ratio to prenatal MBSR or usual care.

Implications for perinatal mental health Teaching the skills of mindfulness meditation to a psychosocially vulnerable group of pregnant women could prove a viable and non-pharmacological approach to improve mental health during pregnancy, reduce stress and support the transition to parenthood. The MBSR program does not target a particular group, and results from the study is thus of potential relevance for pregnant women in general as a means of reducing stress and improving perinatal mental health.

ELIGIBILITY:
Inclusion Criteria:

* Estimated due date no sooner than three months from start of the intervention. This criterion is included in order for the women to be able to complete the intervention before their due date.
* Eighteen + years of age.
* Speak and write Danish.
* Available for group intervention scheduled sessions. Being unavailable for two or more sessions is reason for exclusion from study participation.
* Written informed consent to study criteria.

Exclusion Criteria:

* Active substance dependence.
* Psychotic disorders (e.g. schizophrenia or bipolar disorder).
* Suicidality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The World Health Organization - Five Well-Being Index (WHO-5) | From baseline to 6 months after completion of the intervention.
  The WHO-5 is a global rating scale measuring subjective well-being and consists of five statements and the respondent is asked to rate how well each of the statements applies to her when considering the last 14 days. Each item is scored from 5 "all of the time" to 0 "none of the time". Final scores range from 0 - 100 with higher scores representing greater well-being.

SECONDARY OUTCOMES:
The Depression Anxiety Stress Scales (DASS-21) | From baseline to 6 months after completion of the intervention.
  DASS-21 has three sub-scales designed to discriminate between depression, anxiety and stress in the last week. Each sub-scale include seven items. Response to each item is rated on a four-point Likert scale ranging from 'never' to 'very much/most of the time'. Scores are calculated for each sub-scale and higher scores point to more symptoms of stress, anxiety or depression.
The Edinburgh Depression Scale (EDS) | From baseline to 6 months after completion of the intervention.
  The EDS is a screening questionnaire for depression in the perinatal period that contains 10 questions on how the respondent has felt in the past seven days with each item scored 0 - 3 yielding a maximum score of 30. A higher score points to more depressive symptoms.
The Five-Facet Mindfulness Questionnaire (FFMQ) | From baseline to 6 months after completion of the intervention.
  The FFMQ assesses five general facets of being mindful in daily life: observing, describing, acting with awareness, non-reactivity to inner experience, and non-judging of inner experience. Items are rated on a five-point Likert scale ranging from 1 "never or very rarely true" to 5 "very often or always true". Higher scores suggest higher levels of mindfulness.
The Self-Compassion Scale (SCS) | From baseline to 6 months after completion of the intervention.
  The SCS measures the ability to have a healthy stand towards oneself that does not involve evaluations of self-worth. The scale consists of 12 items and responses are given on a 5-point scale from ranging from 1 "almost never" to 5 "almost always". Higher scores indicate more self-compassionate behavior.

OTHER OUTCOMES:
The Maternal Antenatal Attachment Scale (MAAS) | From baseline to completion of the intervention.
  MASS is a measure of the maternal-fetal bond that consists of 19 items covering two sub-scales: "quality of attachment" (11 items) and "time spent in attachment mode" (8 items) 53. All items are scored on a five-point scale. The minimum score for the total MAAS is 19 and the maximum is 95. The scores for the sub-scales range between 11 and 50 (Quality of attachment) and between 8 and 40 (Time spent in attachment mode). High scores reflect, respectively, a positive quality of attachment and a high intensity of preoccupation with the fetus.
The Childbirth Experience Questionnaire (CEQ) | At 3 months after completion of the intervention.
  The CEQ assess different aspects of childbirth experience 56. The CEQ contains 22 statements assessing four domains of the childbirth experience; own capacity, professional support, participation, and perceived safety. For 19 of the items the response format is a 4-point Likert scale whereas the last three items use a visual analogue scale (VAS). Higher scores reflect a more positive birth experience.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Hvidovre, Copenhagen, Capital Region
  - The Danish Center for Mindfulness, Department of Clinical Medicine, Aarhus University, Aarhus C

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skovbjerg S, Sumbundu A, Kolls M, Kjaerbye-Thygesen A, Fjorback LO. The effect of an adapted Mindfulness-Based Stress Reduction program on mental health, maternal bonding and birth outcomes in psychosocially vulnerable pregnant women: a study protocol for a randomized controlled trial in a Danish hospital-based outpatient setting. BMC Complement Med Ther. 2023 Oct 14;23(1):364. doi: 10.1186/s12906-023-04194-3. PMID 37838672